CLINICAL TRIAL: NCT06161558
Title: Phase 1 Umbrella Trial of Erlotinib In Combination With Select Tyrosine Kinase Inhibitors In Adult Patients With Advanced Solid Tumors
Brief Title: Erlotinib in Combination With Select Tyrosine Kinase Inhibitors in Adult Patients With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of resources to complete study objectives. No participants enrolled.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001657; 001657-C
Record Dates: First submitted 2023-12-07; First posted 2023-12-08 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Neoplasms
Keywords: Kinase Inhibitor; Combination; Pharmacodynamic; TKI
MeSH Terms: conditions — Neoplasms | interventions — Erlotinib Hydrochloride; lenvatinib; Axitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Erlotinib with lenvatinib combination
  Interventions: Drug: Erlotinib; Drug: Lenvatinib
- B (Experimental): Erlotinib with axitinib combination
  Interventions: Drug: Erlotinib; Drug: Axitinib

INTERVENTIONS:
Drug: Erlotinib — Small-molecule tyrosine kinase inhibitor targeting EGFR
Drug: Lenvatinib — Small-molecule tyrosine kinase inhibitor targeting VEGFR1, VEGFR2, and VEGFR3
  Arms: A
Drug: Axitinib — Small-molecule tyrosine kinase inhibitor targeting VEGFR1, VEGFR2, and VEGFR3
  Arms: B

SUMMARY:
Cancers that return or spread after their first line of treatment are often difficult to treat with limited next step options. Based on preclinical studies, the EGFR-targeting tyrosine kinase inhibitor (TKI) Erlotinib may be better in stopping or slowing the growth of tumors when given in combination with the multitargeting TKI Lenvatinib or Axitinib. Participants will be screened with a physical exam and tests including urine and blood tests, imaging scans, and a test of their heart function. Erlotinib, axitinib, and lenvatinib are all capsules taken by mouth. All participants will take their drugs at home every day. Some participants will take erlotinib plus lenvatinib once a day. Some participants will take erlotinib once a day and axitinib twice a day. Assignment to one of the treatment arms will be determined by the study. Participants will record their doses in a diary. Treatment is given in 28-day cycles. All participants will have 4 clinic visits during their first treatment cycle. After that, they will have a clinic visit at the start of each new cycle. Imaging scans, blood and urine tests, and other tests will be repeated during various clinic visits. Participants will remain in the study for as long as the treatment is helping them. They will have follow-up phone calls after they stop treatment....

DETAILED DESCRIPTION:
Primary Objective:

-To establish the safety, tolerability, and maximum tolerated dose (MTD) of the erlotinib-lenvatinib and erlotinib-axitinib combinations in adult patients with advanced solid tumors

Secondary Objective:

-To evaluate the plasma pharmacokinetic profiles of erlotinib and either lenvatinib or axitinib when used in combination

Exploratory Objectives:

* To assess the preliminary antitumor activity of the erlotinib-lenvatinib and erlotinib-axitinib combinations in patients with advanced solid tumors
* To examine changes in numbers of circulating tumor cells (CTCs) of epithelial (cytokeratin+) or mesenchymal (vimentin+) phenotype in response to the erlotinib-lenvatinib or erlotinib-axitinib combinations
* To examine genomic alterations in circulating tumor DNA (ctDNA) that may be associated with response or resistance to the erlotinib-lenvatinib or erlotinib-axitinib combination

Study Design:

* This is an open-label, 2-arm phase 1 trial.
* All agents will be administered orally in 28-day cycles. Dose escalation on both arms will follow a 3 plus 3 design, with intrapatient dose escalation permitted.
* Assignment to one of the treatment arms will be determined by the study.
* The study will allow accrual of patients to backfill cohorts, in which patients will be enrolled on the most recently cleared dose level when accrual to the current dose level has been completed per 3 plus 3 design, but the DLT monitoring period has yet to be completed at that dose level. Dose-limiting toxicities will be defined during the first cycle of treatment.
* The accrual ceiling will be set at 70 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed solid tumors that have progressed on standard therapy known to prolong survival or for which no standard treatment options exist.
* Age >=18 years.
* Patients must have evaluable disease according to RECIST 1.1 criteria.
* ECOG performance status =< 2.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count >=1,500/mcL
  * Platelets >=100,000/mcL
  * Total bilirubin <=1.5 X institutional ULN (with the exception of those with Gilbert syndrome, who must have total bilirubin <=3 X institutional ULN
  * AST(SGOT)/ALT(SGPT) <=3 X institutional upper limit of normal; <= 5.0 x ULN in patients with liver metastases
  * creatinine <=1.5 X institutional ULN

OR

* creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels >1.5 mg/dL

  * Based on preclinical safety data and their respective mechanisms of action, erlotinib, lenvatinib, and axitinib can cause fetal harm when administered to pregnant women. For this reason, women of child-bearing potential and men enrolled on this protocol must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 1 month after dosing with study drugs ceases. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * Potential trial participants should have recovered from clinically significant adverse events of their most recent therapy/intervention prior to enrollment.
  * Patients with non-healing wounds/fistulas may enroll if no immediate surgical input is required in the opinion of the PI.
  * Patients must have <= 1+ proteinuria on urinalysis, or < 1 g protein on 24-hour urine collection, or a urine protein:creatinine ratio of < 1.
  * Prior anti-EGFR- and anti-VEGF/VEGFR-targeted therapy is permitted, provided that the patient has not undergone prior anti-EGFR/anti-VEGF(R) TKI combination therapy.
  * Patients must be able to swallow.
  * Patients with treated brain metastases are eligible if follow-up brain imaging after CNS-directed therapy shows no evidence of progression.
  * Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
  * Patients known to be positive for HIV who meet the following criteria will be considered eligible:
* CD4 count > 350 cells/mm^3
* Undetectable viral load for 6 months prior to enrollment
* Maintained on modern therapeutic regimens utilizing non-CYP-interactive agents
* No history of AIDS-defining opportunistic infections

  * Patients must be willing to provide blood for research purposes.

EXCLUSION CRITERIA:

* For the erlotinib-lenvatinib arm only: patients with a QTcF interval of >=480 msec at study entry or with congenital long QT syndrome are excluded.
* Patients who are receiving any investigational agents are excluded.
* Patients who are receiving >2 anti-hypertensive agents will be excluded.
* Patients who are receiving strong CYP3A4- and/or CYP1A2-inhibiting or -inducing agents that cannot be discontinued or replaced with an alternative medication will be excluded.
* Patients who are receiving agents that increase gastric pH and that cannot be discontinued or replaced with an alternative medication will be excluded.
* Patients who smoke tobacco will be excluded.
* Patients with a history of cirrhosis will be excluded if found to have a moderate or severe Child-Pugh score.
* Patients should not, in the opinion of the Principal Investigator, have GI impairment that may limit the absorption of erlotinib, lenvatinib, or axitinib.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs.
* Uncontrolled intercurrent illness that would, in the opinion of the Principal Investigator, limit compliance with study requirements.
* Pregnant and breastfeeding women are excluded from this study because all 3 study drugs can cause fetal harm, based on preclinical safety data and the respective drug mechanisms of action. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drugs, breastfeeding should be discontinued prior to the first dose of study drug, and women should refrain from nursing throughout the treatment period and for 1 month following the last dose of study drug.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
To establish the safety, tolerability, and maximum tolerated dose (MTD) of the erlotinib-lenvatinib and erlotinib-axitinib combinations in adult patients with advanced solid tumors | 30 months
  This is an open-label phase 1 umbrella trial with 2 treatment arms. All agents will be administered orally in 28-day cycles. The starting dose level (DL) will be DL 1A for Arm A (the erlotinib-lenvatinib combination arm) and DL 1B for Arm B (the erlotinib-axitinib combination arm). Dose escalation on both arms will follow a 3+3 design. Intrapatient dose escalation to the next highest cleared dose level will be permitted upon completion of >= 1 cycle of therapy at the current dose level at which the patient is being treated. Dose-limiting toxicities will be defined during the first cycle of treatment. Patients will be assigned to one of the two treatment arms in an alternating fashion.

SECONDARY OUTCOMES:
To evaluate the plasma pharmacokinetic profiles of erlotinib and either lenvatinib or axitinib when used in combination | 30 months
  Mandatory blood specimens for pharmacokinetic (PK) analysis will be collected aseptically by venipuncture or an existing venous port at baseline and several on-treatment timepoints. Samples will be analyzed using a validated LC-MS/MS method in human plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Shin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Requests for all collected IPD data from clinical trials, conducted under a binding collaborative agreement between NCI/DCTD and a pharmaceutical/biotechnology company, that are not under DSMB monitoring must be in compliance with the terms of the binding collaborative agreement and must be approved by NCI /DCTD and any Pharmaceutical Collaborator.

REFERENCES:
- [Background] Kummar S, Chen HX, Wright J, Holbeck S, Millin MD, Tomaszewski J, Zweibel J, Collins J, Doroshow JH. Utilizing targeted cancer therapeutic agents in combination: novel approaches and urgent requirements. Nat Rev Drug Discov. 2010 Nov;9(11):843-56. doi: 10.1038/nrd3216. Epub 2010 Oct 29. PMID 21031001
- [Background] Conradt L, Godl K, Schaab C, Tebbe A, Eser S, Diersch S, Michalski CW, Kleeff J, Schnieke A, Schmid RM, Saur D, Schneider G. Disclosure of erlotinib as a multikinase inhibitor in pancreatic ductal adenocarcinoma. Neoplasia. 2011 Nov;13(11):1026-34. doi: 10.1593/neo.111016. PMID 22131878
- [Background] Augustin A, Lamerz J, Meistermann H, Golling S, Scheiblich S, Hermann JC, Duchateau-Nguyen G, Tzouros M, Avila DW, Langen H, Essioux L, Klughammer B. Quantitative chemical proteomics profiling differentiates erlotinib from gefitinib in EGFR wild-type non-small cell lung carcinoma cell lines. Mol Cancer Ther. 2013 Apr;12(4):520-9. doi: 10.1158/1535-7163.MCT-12-0880. Epub 2013 Jan 31. PMID 23371860
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001657-C.html